CLINICAL TRIAL: NCT07039773
Title: Assessing Immune Responses to Gluten: A Comparative Study of Liquid Versus Solid Gluten Administration
Brief Title: Gluten Challenge in Celiac Disease - Which Formulation of Gluten Gives the Best Response?
Acronym: SHAKE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Oslo University Hospital (Other)
Collaborators: Lovisenberg (Unknown)
Responsible Party: Principal Investigator, Knut E. A. Lundin, Senior consultant, professor, Oslo University Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 24/27476
Record Dates: First submitted 2025-06-18; First posted 2025-06-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Celiac Disease
Keywords: Gluten challenge; Interleukin-2; Shake; Cookie; T cells; Whole blood cytokine release assay; GI Symptoms
MeSH Terms: conditions — Celiac Disease; Tremor

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten shake (Active Comparator): Liquid form
  Interventions: Dietary Supplement: Vital wheat gluten
- Gluten cookie (Active Comparator): Solid form
  Interventions: Dietary Supplement: Vital wheat gluten

INTERVENTIONS:
Dietary Supplement: Vital wheat gluten — Gluten-containing shake vs gluten-containing cookie
Dietary Supplement: Vital wheat gluten — Half of participants will receive gluten-containing shake first, then gluten-containing cookie next, and vice versa

SUMMARY:
The goal of this clinical trial is to evaluate the immune response to gluten in patients with celiac disease (CeD) by comparing different forms of gluten administration. The participant population includes adults diagnosed with CeD, who are adhering to a gluten-free diet (GFD). The main questions it aims to answer are:

* Does liquid gluten administration elicit a higher IL-2 cytokine response compared to solid gluten administration?
* What is the relationship between serum IL-2 levels and gluten peptide serum concentrations following gluten challenges?

Researchers will compare the responses of two groups: participants receiving liquid gluten (shake) to those receiving solid gluten (cookie) to determine if there is a significant difference in the IL-2 response rates between the two forms.

Participants will be asked to:

* Undergo two gluten challenges (liquid and solid) in a randomized order with at least 4 weeks apart.
* Provide blood samples before and after each challenge to measure serum IL-2 levels and gluten peptide concentrations over a period of 6 hours.
* Report any symptoms experienced following each gluten challenge.

ELIGIBILITY:
Inclusion Criteria:

* BMI 18-33 kg/m2
* Willingness to comply with the study procedure and having signed informed, written consent
* Previous diagnosis of coeliac disease according to established guidelines based on positive serology (Endomysium test, IgA-TG2 and/or IgG-DGP) (diagnosed in childhood) and a duodenal biopsy showing villous atrophy graded as Marsh 3 according to guidelines from European Society for Study of Coeliac Disease .
* Strict adherence to a gluten-free diet at least the 12 last months.

Exclusion Criteria:

* Positive serology (IgA-TG2 below upper level of normal) at screening visit
* Pregnancy or breast feeding. Fertile women must use effective contraception.
* Other inflammatory disease like uncontrolled hypothyreosis, type 1 diabetes, cardiovascular diseases, thyroid and renal disorders, inflammatory bowel diseases or any other disease that in the opinion of the responsible clinician makes the patient unsuitable for the study
* Using of immunosuppressive/steroid medications
* Wheat allergy
* Severe acute infection

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Comparison of serum IL-2 response rates between the gluten shake group and the cookie group | From baseline to 4 hours at visit 1
  A responder is defined as an individual exhibiting a log-transformed cytokine level equal to or greater than 0. This level corresponds to 1.0 pg/ml in concentration of IL-2 in serum. The hypothesis is that there is a higher proportion of responders in the gluten shake group compared to the cookie group.

SECONDARY OUTCOMES:
Correlation between serum IL-2 response levels and baseline whole blood plasma IL-2 | From baseline to 6 hours after gluten intake
Correlation between serum IL-2 response levels and baseline number of gluten-specific T cells | From baseline to 6 hours after gluten intake
Correlation between serum IL-2 response levels and symptom severity | From baseline to 6 hours after gluten intake
Comparison of serum IL-2 response levels and serum gluten peptide levels | From baseline to 6 hours after gluten intake

CONTACTS AND LOCATIONS:
Locations (2):
- Norway (2):
  - Oslo University Hospital, Oslo, Oslo County
  - Lovisenberg Diakonale Hospital, Oslo, Oslo County

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tye-Din JA, Daveson AJM, Goldstein KE, Hand HL, Neff KM, Goel G, Williams LJ, Truitt KE, Anderson RP; RESET CeD Study Group. Patient factors influencing acute gluten reactions and cytokine release in treated coeliac disease. BMC Med. 2020 Nov 26;18(1):362. doi: 10.1186/s12916-020-01828-y. PMID 33239013
- [Background] Goel G, Daveson AJM, Hooi CE, Tye-Din JA, Wang S, Szymczak E, Williams LJ, Dzuris JL, Neff KM, Truitt KE, Anderson RP. Serum cytokines elevated during gluten-mediated cytokine release in coeliac disease. Clin Exp Immunol. 2020 Jan;199(1):68-78. doi: 10.1111/cei.13369. Epub 2019 Oct 1. PMID 31505020